CLINICAL TRIAL: NCT02744183
Title: Training in the Fasted State, Glucose Metabolism and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Dr Javier Gonzalez, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EP 15/16129
Record Dates: First submitted 2016-04-11; First posted 2016-04-20 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Glucose Metabolism Disorders
Keywords: Exercise; Fasted; Glucose; Energy Balance
MeSH Terms: conditions — Glucose Metabolism Disorders; Motor Activity | interventions — Exercise; Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Group (Active Comparator): Maintain habitual habits
  Interventions: Behavioral: Maintain habitual habits
- Fed Exercise (Active Comparator): 6 weeks of moderate intensity exercise with breakfast consumption
  Interventions: Behavioral: Exercise; Behavioral: Breakfast
- Fasted Exercise (Experimental): 6 weeks of moderate intensity exercise with breakfast omission
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Moderate intensity exercise
  Arms: Fasted Exercise; Fed Exercise
Behavioral: Breakfast — Breakfast consumption
  Arms: Fed Exercise
Behavioral: Maintain habitual habits — Normal physical activity and dietary behaviors maintained
  Arms: Control Group

SUMMARY:
In healthy individuals, the body responds to glucose (sugar) ingestion by reducing the amount released from the liver. At the same time, skeletal muscles increase the rate at which they remove the glucose from the bloodstream, via the actions of the hormone insulin. This ensures that blood glucose levels remain in a controlled range. However, in developed countries, diseases such as metabolic syndrome and type 2 diabetes are becoming prevalent, due to dietary modifications and a reduction in physical activity. As one of the prominent barriers to regular physical activity is a lack of time, finding ways to maximize the health benefits of exercise is a priority for researchers.

The investigators want to understand potential differences in the effects of six weeks of aerobic training, with the exercise performed either after breakfast or after a prolonged fast. Specifically, this research aims to investigate whether there is a difference in the change in processes implicated in glucose regulation and secondly, in subsequent eating and physical activity behaviors. By investigating these changes this work will explore how exercise and nutrition can be optimized to benefit health and weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-49
* Body mass index (BMI) > 25 kg/m2
* Weight stable for > 6 months
* Not currently engaging in any form of structured exercise
* Be able and willing to give informed oral and written consent
* Complete and meet the defined criteria of pre-study questionnaires and screen

Exclusion Criteria:

* Have a history of metabolic, cardio-pulmonary or musculoskeletal disease
* Have plans to change diet and/or physical activity outside of the intervention
* Taking regular medication or food supplements from which it is not possible to refrain and which are known to influence any of the outcome measures.
* Failure to refrain from alcohol and/or caffeine containing drinks or strenuous exercise one day before or during the trial days
* Smokers
* Any reported condition or behavior deemed to pose a risk to the participant or introduce bias into the experiment

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma glucose concentrations | 120 mins - (change after 6 weeks)
  Response to oral glucose tolerance test (area under the curve)
Postprandial insulin concentrations | 120 mins - (change after 6 weeks)
  Response to oral glucose tolerance test (area under the curve)

SECONDARY OUTCOMES:
Oral Glucose Insulin Sensitivity Index | 120 mins - (change after 6 weeks)
  Response to oral glucose tolerance test
Cardiorespiratory fitness (VO2max) | Change after 6 weeks
Habitual energy intake | Change after 6 weeks
  Assessed via a food diary, completed at baseline and during the last week of the intervention
Habitual energy expenditure | Change after 6 weeks
  Assessed via an Actiheart monitor, completed at baseline and during the last week of the intervention
Body mass (kg) | Change after 6 weeks
Waist and hip circumference (cm) | Change after 6 weeks
Maximal rate of whole-body lipid oxidation (g/min) | Change after 6 weeks
  During an incremental exercise test
Fasting plasma glucose concentration | Basal Concentrations - (change after 6 weeks)
  Fasting plasma glucose concentration (mmol/L)
Fasting plasma insulin concentration | Basal Concentrations - (change after 6 weeks)
  Fasting plasma insulin concentration (pmol/L)
Postprandial non-esterified fatty acid concentrations | 120 mins - (change after 6 weeks)
  Response to oral glucose tolerance test (total and incremental area under the curve)
Fasting plasma triglyceride concentrations | Basal Concentrations - (change after 6 weeks)
  Fasting plasma triglyceride concentrations (mmol/L)
Fasting plasma total cholesterol concentrations | Basal Concentrations - (change after 6 weeks)
  Fasting plasma total cholesterol concentrations (mmol/L)
Fasting plasma HDL cholesterol concentrations | Basal Concentrations - (change after 6 weeks)
  Fasting plasma HDL cholesterol concentrations (mmol/L)
Fasting plasma LDL cholesterol concentrations | Basal Concentrations - (change after 6 weeks)
  Fasting plasma LDL cholesterol concentrations (mmol/L)
Fasting plasma non-esterified fatty acid concentrations | Basal Concentrations - (change after 6 weeks)
  Fasting plasma non-esterified fatty acid concentrations (mmol/L)
Waist to hip ratio | Change after 6 weeks
  Waist circumference (cm) divided by hip circumference (cm)
Citrate Synthase Activity (mitochondrial citrate synthase activity in each muscle sample in an immunocapture based manner) | Change after 6 weeks
  Skeletal muscle (vastus lateralis). Citrate Synthase Activity Assay Kit.
Protein content of mitochondrial respiratory chain proteins | Change after 6 weeks. For each participant the protein content will be presented as the fold change from baseline (arbitrary units).
  Skeletal muscle (vastus lateralis). Complex I, Complex II, Complex III, Complex IV.
Protein content of carnitine palmitoyltransferase I (CPT-1) | Change after 6 weeks. For each participant the protein content will be presented as the fold change from baseline (arbitrary units)
  Skeletal muscle (vastus lateralis)
Protein content of cluster of differentiation 36 (CD36) | Change after 6 weeks. For each participant the protein content will be presented as the fold change from baseline (arbitrary units)
  Skeletal muscle (vastus lateralis)
Protein content (total and phosphorylated form) of AMP-activated protein kinase (AMPK) | Change after 6 weeks. For each participant the protein content will be presented as the fold change from baseline (arbitrary units)
  Skeletal muscle (vastus lateralis)
Resting metabolic rate (RMR) | Change after 6 weeks
  Assessed via indirect calirometry
Energy balance | Change after 6 weeks (during week 6 of intervention versus baseline monitoring)
  Total energy expenditure minus total energy intake
Whole-body lipid utilisation during exercise | Change throughout complete training period (weeks 1 through to 6). Samples will be collected during every training session (three times weekly for six weeks)
  Assessed via indirect calirometry during every exercise session (at ten minute intervals)
Whole-body carbohydrate utilisation during exercise | Change throughout complete training period (weeks 1 through to 6). Samples will be collected during every training session (three times weekly for six weeks)
  Assessed via indirect calirometry during every exercise session (at ten minute intervals)
Homeostasis Model Assessment (HOMA2-IR) | Change after 6 weeks
  The Homeostasis Model Assessment (HOMA) estimate of steady state beta cell function (%B) and insulin sensitivity (%S). Derived from fasting plasma glucose and fasting plasma insulin concentrations.
Fasting plasma glycerol concentrations | Basal Concentrations - (change after 6 weeks)
  Fasting plasma glycerol concentrations (mmol/L)
Postprandial plasma glycerol concentrations | Change after 6 weeks
  Response to oral glucose tolerance test (total and incremental area under the curve)
Adipose Tissue Insulin Resistance Index (Adipo-IR) | Change after 6 weeks
  Response to oral glucose tolerance test (total and incremental area under the curve)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Gonzalez, PhD, Principal Investigator — University of Bath
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonzalez JT, Veasey RC, Rumbold PL, Stevenson EJ. Breakfast and exercise contingently affect postprandial metabolism and energy balance in physically active males. Br J Nutr. 2013 Aug;110(4):721-32. doi: 10.1017/S0007114512005582. Epub 2013 Jan 29. PMID 23340006
- [Background] Van Proeyen K, Szlufcik K, Nielens H, Pelgrim K, Deldicque L, Hesselink M, Van Veldhoven PP, Hespel P. Training in the fasted state improves glucose tolerance during fat-rich diet. J Physiol. 2010 Nov 1;588(Pt 21):4289-302. doi: 10.1113/jphysiol.2010.196493. PMID 20837645
- [Derived] Edinburgh RM, Bradley HE, Abdullah NF, Robinson SL, Chrzanowski-Smith OJ, Walhin JP, Joanisse S, Manolopoulos KN, Philp A, Hengist A, Chabowski A, Brodsky FM, Koumanov F, Betts JA, Thompson D, Wallis GA, Gonzalez JT. Lipid Metabolism Links Nutrient-Exercise Timing to Insulin Sensitivity in Men Classified as Overweight or Obese. J Clin Endocrinol Metab. 2020 Mar 1;105(3):660-76. doi: 10.1210/clinem/dgz104. PMID 31628477